CLINICAL TRIAL: NCT02759731
Title: A Phase 1/2 Study of Baricitinib, a JAK1/2 Inhibitor, in Chronic Graft-Versus-Host Disease (cGVHD) After Allogeneic Hematopoietic Stem Cell Transplantation (SCT)
Brief Title: Study of Baricitinib, a JAK1/2 Inhibitor, in Chronic Graft-Versus-Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Pavletic, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160094; 16-C-0094
Record Dates: First submitted 2016-04-14; First posted 2016-05-03 (Estimated); Results first posted 2023-10-25 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Graft vs Host Disease; Chronic Graft-Versus-Host Disease
Keywords: Murine Models; Rheumatoid Arthritis; Corticosteroids; Systemic Therapy; Inflammatory Cytokines
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Single arm, intra-patient dose escalation. Arm 1 (starting dose) -Baricitinib starting at a dose of 2mg daily for 12 weeks. If the response at 12 weeks is a complete response (CR) and there has not been a dose-limiting toxicity (DLT), the dose will remain at 2mg daily for an additional 12 weeks. Arm 2 (dose escalation) - If the response is a partial response (PR) or stable disease (from cohort 1), the dose will be increased to 4mg daily for an additional 12 weeks. If there has been a DLT within the first 4 weeks will have a dose reduction back to 2mg daily.
  Each participant is exposed to both dose levels (with the exception of participants who developed toxicity or progressive disease that caused them to discontinue study early before they were able to undergo the per-protocol dose escalation at 12 weeks).
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Cycle=28 days: Baricitinib: 1mg-4mg by mouth (PO) every day (QD)
  Other Names: Olumiant

SUMMARY:
Background:

Chronic graft versus host disease (cGVHD) can affect people who had a hematopoietic stem cell transplant using donor cells. It is often fatal. It is usually treated with high doses of steroids. But that helps only about half the people in the long term. Researchers want to see if a drug called baricitinib can help people with cGVHD that has not responded to therapy. The drug inhibits the proteins involved in communication in the immune system. These proteins may play a role in cGVHD and other inflammatory diseases.

Objectives:

To test the safety and effectiveness of baricitinib in people with cGVHD that has not responded to therapy.

Eligibility:

Adults 18 and older with cGVHD that has not responded to therapy.

Design:

Participants will be screened with a medical history, physical exam, and blood and urine tests. They will have lung and heart tests and chest scans.

Baseline visit: Participants will have:

Medical history

Physical exam

Blood tests

Tests for infectious diseases

Skin, eye, and teeth evaluations

Rehabilitation and occupational medicine evaluations

Photos of any lesions

Gynecology evaluation (females)

The study will occur in 28-day cycles. Participants will take the study drug by mouth every day for 3 cycles. Some will take it for 3 or 6 more cycles.

Participants will have a few visits during each cycle. They will repeat some previous tests. They may also have scans and questionnaires.

Participants will have a visit when they stop taking the drug and another 3 months later. They will repeat a few study tests. They will have follow-up calls for 2 years.

DETAILED DESCRIPTION:
* Background:

  * Chronic graft-versus-host disease (cGVHD) is the leading cause of non-relapse morbidity and mortality in persons after allogeneic hematopoietic stem cell transplantation (SCT).
  * Approximately 50% of patients with cGVHD have disease refractory to systemic corticosteroids; currently, there is no standard second-line therapy.
  * The Janus kinase/signal transducers and activators of transcription (JAK/STAT) pathway relays the signaling function of several inflammatory cytokines that have a role in GVHD (interferon (IFN)-gamma, Interleukin-2 (IL-2), Interleukin-6 (IL-6), Interleukin-12 (IL-12)).
  * Murine models have demonstrated activity of JAK inhibitors in graft-versus-host disease.
  * Baricitinib is a potent and selective inhibitor of Janus kinase 1 (JAK1) and Janus kinase 1 (JAK2) that has demonstrated anti-inflammatory effects and a good safety profile in patients with rheumatoid arthritis but has not been evaluated in GVHD.
* Objectives:

  * To determine the safety and tolerability of baricitinib in patients with cGVHD that is refractory to steroids
  * To determine the efficacy of baricitinib in patients with cGVHD that is refractory to steroids
* Eligibility:

  * Inclusion:

    * Age greater than or equal to 18 years
    * Moderate or severe cGVHD per NIH consensus criteria
    * Karnofsky performance status greater than or equal to 50%
    * cGVHD that did not respond to high-dose corticosteroids (prednisone at 1.0 mg/kg/day for at least 1 week or prednisone at 0.5 mg/kg/day or 1 mg/kg every other day for at least 4 weeks), or second-line therapy (any)
    * Receiving stable or tapering doses of systemic therapy in the preceding 4 weeks if taking systemic therapy for cGVHD
  * Exclusion:

    * Neutrophils <1.0x10^9/L, platelets <50X10^9/L, creatinine greater than or equal to 1.5 times the upper limit of normal or estimated creatinine clearance <50mL/min/1.73m^2 (Cockroft-Gault formula), serum aspartate aminotransferase or alanine aminotransferase concentration >3x upper limit of normal (ULN) or total bilirubin greater than or equal to 1.5x ULN
    * Progressive malignancy, uncontrolled infection or any major organ dysfunction as defined by the protocol
* Design:

  * This is a Phase 1/2 trial to determine the safety and efficacy of baricitinib in patients with cGVHD that is refractory to steroids.
  * Patients will initially be treated with baricitinib at 2mg daily for 12 weeks. If the response at 12 weeks is a complete response (CR) and there has not been a dose-limiting toxicity (DLT), the dose will remain at 2mg daily for an additional 12 weeks, with the primary response assessment at 24 weeks of total treatment. If the response is a partial response (PR) or stable disease, the dose will be increased to 4mg daily for an additional 12 weeks, with the primary response assessment at 24 weeks of total treatment. If there is progression of disease at any time within the first 12 weeks, the dose can be increased to 4mg daily at that time, and patients will continue for a total of 24 weeks of treatment. Patients will have the option to continue baricitinib for an additional 6 months as tolerated if they have stable or responding disease.
  * The co-primary endpoint of safety will be determined by rate, severity, and duration of adverse events based on Common Terminology Criteria for Adverse Events (CTCAE) v4 criteria. Assessment for DLTs will occur every 2 weeks during the first 4 weeks of each dose level. Safety monitoring will occur every 4 weeks thereafter.
  * The co-primary endpoint of efficacy will be defined as rate of overall response at 24 weeks per National Institutes of Health (NIH) consensus criteria (CR or PR).
  * Peripheral blood samples will be collected prior to treatment, at 2 weeks, at 12 weeks and every 12 weeks thereafter to evaluate cytokine and cellular profiles, STAT phosphorylation, candidate chronic GVHD biomarkers. Pharmacokinetic studies will also be performed at each dose level.
  * In an initial futility analysis, if 0 of the first 7 patients enrolled in cohort 1 have responded at 12 weeks, then a 2nd cohort of patients will be accrued to start treatment at the higher dose (4mg daily). Otherwise, if 1 or more of the first 7 patients respond in cohort 1, then 21 evaluable patients will be treated in cohort 1. Similarly, if the second cohort is used, and if 0 of the 7 patients enrolled in this second cohort have responded at 12 weeks, then no further patients will be accrued. Otherwise, if 1 or more of the first 7 patients respond in cohort 2, then 21 evaluable patients will be treated in cohort 2.
  * A total of 21 evaluable patients will be enrolled in either cohort 1 or 2 as appropriate, in order to have 80% power to detect a response rate consistent with 30% and ruling out 10%, with a one-sided significance level of 0.10 for the cohort. As an early stopping rule for safety, if 2/3 or greater patients at any given dose level experiences a dose limiting toxicity requiring dose reduction or discontinuation, that dose will not be subsequently used, and no further dose escalation will take place.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Moderate or severe Chronic Graft-Versus-Host Disease (cGVHD) (after allogeneic hematopoietic stem cell transplantation) diagnosed and staged per National Institutes of Health (NIH) criteria. Responses to Janus kinase (JAK) inhibitors have not been restricted to specific organs, so any organ involvement is eligible.
2. Age greater than or equal to 18 years of age. Because inadequate dosing or adverse event data are currently available on the use of baricitinib in patients <18 years of age, children are excluded from this study.
3. Karnofsky performance score >50%
4. Chronic GVHD that did not respond to high-dose corticosteroids (prednisone at 1.0 mg/kg/day for at least 1 week or prednisone at 0.5 mg/kg/day or 1 mg/kg every other day for at least 4 weeks), or second-line therapy (any).
5. If patient is taking systemic therapy for cGVHD at the time of enrollment, they must be on a stable or tapering doses in the preceding 4 weeks.
6. Patients must have normal organ and marrow function as defined below:

   absolute neutrophil count greater than or equal to 1,000/mcL

   absolute lymphocyte count greater than or equal to 500/mcL

   platelets greater than or equal to 50,000/mcL

   hemoglobin greater than or equal to 9 g/dL

   total bilirubin less than or equal to 1.5 X institutional upper limit of normal, unless there is a known history of Gilbert's disease

   Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) serum glutamic pyruvic transferase (SGPT) less than or equal to 3 X institutional upper limit of normal
   * Creatinine < 1.5 times the upper limit of normal, or:

   creatinine clearance greater than or equal to 50 mL/min/1.73 m^2. Creatinine clearance should be calculated per institutional standard.
7. Primary malignancy for which the patient received transplant has been stable for 3 months prior to enrollment on study.
8. The effects of baricitinib on human fetal development are unknown. Women of child-bearing potential and men must agree to use 2 effective forms of contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for at least 7 days after study drug exposure. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, or if a man's partner becomes pregnant or suspects she is pregnant while he is participating in this study, she or he should inform their treating physician immediately.
9. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Systemic immune suppression or systemic therapy for cGVHD started within preceding 4 weeks.
2. Hypersensitivity to JAK inhibitors.
3. Any serious medical condition within the previous 4 weeks which places the subject at an unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study, including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmias, acute kidney injury, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Uncontrolled infection, including active human immunodeficiency virus (HIV-1), Hepatitis B virus (HBV) and/or Hepatitis C virus (HCV) infection (positive HBV or HCV viral load in the setting of positive HBV core antibody or surface antibody or HCV antibody). History of HBV or HCV is allowed if there is no uncontrolled viral infection. Because the study agent may impact response to infections, patients with any active viral infection are excluded.
5. Recurrent or progressive malignancy requiring anticancer treatment.
6. Other cancer except that for which the transplant was done <2 years before study entry, except non-melanoma skin cancer or carcinoma in situ of the uterine cervix or breast.
7. Patients who are receiving any other investigational agents.
8. NIH lung score 3.
9. Pregnant women are excluded from this study because the teratogenic effects of baricitinib are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with baricitinib, breastfeeding should be discontinued if the mother is treated with this agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0094.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single arm study (with intra-patient dose escalation) - so all participants are exposed to both dose levels unless they prematurely developed toxicity that led to study discontinuation or dose modification. We report as one arm and then report the dose modifications/discontinuation separately - but the modification/discontinuation does not define those participants as a separate group.
Groups:
- Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib: Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib
Period: Overall Study
Arm/Group | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib
Started | 24
Completed | 16
Not Completed | 8
Not completed — Did not complete treatment. | 8

BASELINE CHARACTERISTICS:
Population: This is a single arm study (with intra-patient dose escalation) - so all participants are exposed to both dose levels unless they prematurely developed toxicity that led to study discontinuation or dose modification. We report as one arm and then report the dose modifications/discontinuation separately - but the modification/discontinuation does not define those participants as a separate group.
Arm/Group | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLT is defined as any grade ≥3 non-hematologic or grade ≥4 hematologic adverse event, or hemoglobin <6.5 g/dL, within 4 weeks of starting any dose level (1mg, 2mg, or 4 mg) except those that are clearly and incontrovertibly due to extraneous causes. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: Starting at each dose level initiation, every 2 weeks up to the first 4 weeks of each dose
Population: Single arm study (intra-patient(pt) dose escalation). All pts exposed to both dose levels(DL) unless prematurely developed toxicity that led to study discontinuation/dose modification. We report as 1 arm&then report dose modifications/discontinuation separately. Modification/discontinuation does not define those pts as a separate group. 20/24pts analyzed DL2 because they never made it to 3month mark when dose escalation occurred/never underwent dose escalation to 4mg due to toxicity/progression.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1, 2 mg of Baricitinib: Dose Level 1, 2 mg of Baricitinib
- Dose Level 2, 4 mg of Baricitinib: Dose Level 2, 4 mg of Baricitinib
Arm/Group | Dose Level 1, 2 mg of Baricitinib | Dose Level 2, 4 mg of Baricitinib
Number analyzed (Participants) | 24 | 20
Participants | 0 | 0

2. Primary Outcome: Phase 2: Number of Participants With Any Serious and/or Non-Serious Grades 3, 4, and/or 5 Adverse Events Due to Drug
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 3 is severe. Grade 4 is life-threatening. And Grade 5 is death related to adverse event.
Time Frame: every 4 weeks through study completion (up to 48 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib
Number analyzed (Participants) | 24
Participants
  Grade 3 | 2
  Grade 4 | 0
  Grade 5 | 0

3. Primary Outcome: Phase 2: Overall Response at 24 Weeks
Description: Response was assessed by the National Institutes of Health (NIH) chronic graft-versus-host disease (cGVHD) response criteria. Complete Response (CR) is defined as resolution of all manifestations in each organ or site. Partial Response (PR) is defined as improvement at least 1 organ or site without progression in any other organ or site. Lack of Response including unchanged, mixed response, and disease progression. Mixed response is a CR or PR in at least 1 organ accompanied by progression in another organ. Unchanged is outcomes that do not meet the criteria for CR, PR, disease progression, or mixed response. Disease Progression is a change in the manifestations in each organ or site that does not meet the criteria for CR, PR, mixed response, unchanged or lack of response.
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib
Number analyzed (Participants) | 24
Participants
  Complete Response | 0
  Partial Response | 16
  Mixed Response | 3
  Unchanged | 0
  Disease Progression | 0
  Not Evaluable: participants did not make it to the 24-week mark for response assessment. | 5

4. Other Pre Specified Outcome: Phase 1 and 2: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to 30 days off study drug, approximately 73 months and 28 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib
Number analyzed (Participants) | 24
Participants | 21

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to 30 days off study drug, approximately 73 months and 28 days.
Description: Single arm study (intra-patient (pt) dose escalation). All pts is exposed to both dose levels unless prematurely developed toxicity that led to study discontinuation/dose modification. We report as 1 arm&then report dose modifications/discontinuation separately. The modification/discontinuation does not define those pts as a separate group. We cannot report adverse events(AEs) per dose level as some late AEs are considered cumulative from exposure to drug which was interchangeable and increased.
Arm/Group | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 8/24
Other Adverse Events (participants affected / at risk) | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib (N=24)
Anaphylaxis (Immune system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, Post transplant lymphoproliferative disorder (Blood and lymphatic system disorders) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Bone infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1, 2 mg of Baricitinib -> Dose Level 2, 4 mg of Baricitinib (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, Lymphadenopathy (CT) (Blood and lymphatic system disorders) | 1 (1)
Carbon monoxide diffusing capacity decreased (Investigations) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Cholesterol high (Investigations) | 2 (3)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2)
Eye disorders - Other, Chalazion RUL (Eye disorders) | 1 (1)
Eye infection (Infections and infestations) | 1 (2)
Eye pain (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Forced expiratory volume decreased (Investigations) | 3 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (8)
Hypotension (Vascular disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, Sputum culture + for Pseudomonas a. (Infections and infestations) | 1 (1)
Infections and infestations - Other, Thrush (Infections and infestations) | 1 (1)
Infections and infestations - Other, scabies (Infections and infestations) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, Right peroneus brevis tendon tear (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, srt. wrist sprain (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Lung infection (Infections and infestations) | 3 (4)
Lymphocyte count decreased (Investigations) | 2 (4)
Metabolism and nutrition disorders - Other, metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, muscle spasms, pain and stiffness upper arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Other, Carcinoma in situ of lower lip
Neutrophil count decreased (Investigations) | 2 (6)
Otitis externa (Ear and labyrinth disorders) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Oral pyogenic granuloma (Skin and subcutaneous tissue disorders) | 1 (2)
Skin infection (Infections and infestations) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 8 (14)
Vomiting (Gastrointestinal disorders) | 1 (2)
Weight gain (Investigations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02759731/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT02759731/ICF_001.pdf